CLINICAL TRIAL: NCT02477891
Title: An Open-Label Treatment Use Protocol for Daratumumab in Subjects With Multiple Myeloma Who Have Received at Least 3 Prior Lines of Therapy (Including a Proteasome Inhibitor and an Immunomodulatory Agent) or Are Double Refractory to a Proteasome Inhibitor and an Immunomodulatory Agent
Brief Title: Early Access Treatment With Daratumumab for (Relapsed or Refractory) Multiple Myeloma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106626; 54767414MMY3010 (Other: Janssen Research & Development, LLC); 2015-002993-19 (EudraCT Number)
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Daratumumab; Early access
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Daratumumab — Participants will receive daratumumab (16 milligram per kilogram [mg/kg]) as intravenous infusion on Day 1, 8, 15, and 22 of Cycles 1 and 2 (weekly dosing), on Day 1 and 15 of Cycles 3 to 6 (every 2 weeks dosing), and on Day 1 of Cycle 7 and subsequent cycles (every 4 weeks dosing) until documented progression, unacceptable toxicity, or study end. Each cycle is of 28 days.

SUMMARY:
The objective of this study is to provide early access to daratumumab treatment and collect additional safety data while the medication is not commercially available or available through another protocol for subjects with multiple myeloma who have received at least 3 prior lines of therapy including a proteasome inhibitor (PI) and an immunomodulatory agent (IMiD) or whose disease is double refractory to both a PI and an IMiD.

DETAILED DESCRIPTION:
This is a multicenter, open-label, early access treatment protocol of single-agent daratumumab in subjects with multiple myeloma who have received at least 3 prior lines of therapy including a PI and an IMiD or whose disease is double refractory to both a PI and an IMiD, who reside in areas where daratumumab is not commercially available or available through another protocol, who have not been enrolled in another daratumumab study, and who are not eligible for or who do not have access to enrollment in another ongoing clinical study of daratumumab. The study will have three phases: Screening phase (30 days prior to first dose of study drug), treatment phase (until documented progression, unacceptable toxicity, or study end), End of Treatment (30 days after last dose of study drug). Participants will receive daratumumab (16 milligram per kilogram [mg/kg]) as intravenous infusion. Participants will primarily be assessed for overall response rate. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age
* Subject must have documented multiple myeloma and have evidence of disease progression on or after the most recent prior treatment regimen as defined by IMWG criteria: Subjects who have received at least 3 prior lines of therapy including a proteasome inhibitor (greater than or equal to [>=] 2 cycles or 2 months of treatment) and an IMiD (>= 2 cycles or 2 months of treatment) in any order during the course of treatment (except for subjects who discontinued either of these treatments due to a severe allergic reaction within the first 2 cycles/months) OR Subjects whose disease is double refractory to a proteasome inhibitor (PI) and an immunomodulatory agent (IMiD). For subjects who have received more than 1 type of PI, their disease must be refractory to the most recent one. Similarly, for those who have received more than 1 type of IMiD, their disease must be refractory to the most recent one
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* A woman of childbearing potential must have a negative serum or urine pregnancy test at Screening
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control during the study, and all men must also not donate sperm during the study and for 6 months after receiving the last dose of study drug

Exclusion Criteria:

* Ever enrolled in another daratumumab study or eligible for enrollment in another ongoing clinical study of daratumumab
* Subject receives any other anti-myeloma therapy while receiving daratumumab
* Enrolled in another interventional clinical study with therapeutic intent
* Subject has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) less than 50% of predicted normal
* Subject has known moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification
* Prior exposure to any anti-CD38 monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (79):
- United States (41):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Duarte, California
  - Fountain Valley, California
  - Gilroy, California
  - Greenbrae, California
  - Los Angeles, California
  - West Hollywood, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Ocala, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Topeka, Kansas
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Great Falls, Montana
  - Omaha, Nebraska
  - Flemington, New Jersey
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Buffalo, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Corvallis, Oregon
  - Hershey, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Fairfax, Virginia
- Brazil (6):
  - Barretos
  - João Pessoa
  - Porto Alegre
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Kobe, Japan
- Russia (5):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Samara
  - Volgograd
- Spain (13):
  - Barcelona
  - Granada
  - Las Palmas de Gran Canaria
  - Madrid
  - Mallorca
  - Pamplona
  - Salamanca
  - Santander
  - Santiago de Compostela
  - Toledo
  - Valencia
  - Valladolid
  - Zaragoza
- United Kingdom (13):
  - Blackpool
  - Bournemouth
  - Dundee
  - Glasgow
  - Kent
  - Leeds
  - London
  - Londonderry
  - Manchester
  - Newcastle
  - Nottingham
  - Stoke-on-Trent
  - Wolverhampton

REFERENCES:
- [Derived] Cook G, Corso A, Streetly M, Mendeleeva LP, Ptushkin VV, Chan E, Ukropec J, Iraqi W, Al-Akabawi A, Pei H, Gaudig M, Petrucci MT, Alegre A, Mateos MV. Daratumumab Monotherapy for Relapsed or Refractory Multiple Myeloma: Results of an Early Access Treatment Protocol in Europe and Russia. Oncol Ther. 2021 Jun;9(1):139-151. doi: 10.1007/s40487-020-00137-x. Epub 2021 Feb 25. PMID 33630275
- [Derived] Crusoe EQ, Pimenta FCF, Maiolino A, Castro NS, Pei H, Trufelli D, Fernandez M, Herriot LB. Results of the daratumumab monotherapy early access treatment protocol in patients from Brazil with relapsed or refractory multiple myeloma. Hematol Transfus Cell Ther. 2021 Oct-Dec;43(4):417-423. doi: 10.1016/j.htct.2020.07.005. Epub 2020 Sep 14. PMID 32967807